CLINICAL TRIAL: NCT03901963
Title: A Randomized Study of Daratumumab Plus Lenalidomide Versus Lenalidomide Alone as Maintenance Treatment in Patients With Newly Diagnosed Multiple Myeloma Who Are Minimal Residual Disease Positive After Frontline Autologous Stem Cell Transplant
Brief Title: A Study of Daratumumab Plus Lenalidomide Versus Lenalidomide Alone as Maintenance Treatment in Participants With Newly Diagnosed Multiple Myeloma Who Are Minimal Residual Disease Positive After Frontline Autologous Stem Cell Transplant
Acronym: AURIGA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108599; 54767414MMY3021 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daratumumab + Lenalidomide (Experimental): Participants will receive 1800 milligram (mg) daratumumab by subcutaneous (SC) injection in combination with lenalidomide (orally) as maintenance therapy for a maximum of 36 cycles. Each cycle is of 28 days.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide
- Lenalidomide (Active Comparator): Participants will receive lenalidomide (orally) alone as maintenance therapy for a maximum of 36 cycles. Each cycle is of 28 days.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 1800 mg will be administered by SC injection weekly during Cycles 1 and 2, every 2 weeks during Cycles 3 through 6, and every 4 weeks from Cycle 7 onward until confirmed progressive disease (PD), unacceptable toxicity, or until end of study treatment for a maximum of 36 cycles.
  Other Names: DARZALEX
  Arms: Daratumumab + Lenalidomide
Drug: Lenalidomide — Lenalidomide 10 mg will be administered orally from Day 1 to Day 28 (continuously) of each 28-day cycle until confirmed PD, unacceptable toxicity, or until end of study treatment for a maximum of 36 cycles. After 3 cycles of maintenance therapy, if well tolerated, the lenalidomide dose may be increased to 15 mg daily, at the discretion of the investigator.

SUMMARY:
The purpose of this study is to evaluate conversion rate to minimal residual disease (MRD) negativity following the addition of daratumumab to lenalidomide relative to lenalidomide alone, when administered as maintenance treatment to anti-cluster of differentiation 38 (CD38) treatment naive participants with newly diagnosed multiple myeloma who are MRD positive as determined by next generation sequencing (NGS) at screening, following high-dose therapy (HDT) and autologous stem cell transplant (ASCT).

ELIGIBILITY:
Inclusion Criteria:

* Must have newly diagnosed multiple myeloma with a history of a minimum of 4 cycles of induction therapy, have received high-dose therapy (HDT) and autologous stem cell transplantation (ASCT) within 12 months of the start of induction therapy, and be within 6 months of ASCT on the date of randomization
* Must have a very good partial response (VGPR) or better response assessed per International Myeloma Working Group (IMWG) 2016 criteria at the time of randomization
* Must have archived bone marrow samples collected before induction treatment (that is, at diagnosis) or before transplant (for example, at the end of induction) or have existing results on the index multiple myeloma clone based on Adaptive Biotechnologies' next generation sequencing (NGS)-based minimal residual disease (MRD) assay. Archived bone marrow samples will be used for calibration of myeloma clonal cells to facilitate assessment of primary end point by NGS. If an existing result on index myeloma clone is available from Adaptive Biotechnologies' NGS-based MRD assay, as part of institutional procedures, an archived bone marrow sample is not required as long as Adaptive Biotechnologies is able to retrieve historical results on the index myeloma clone form the clinical database. Any one of the following archived samples are required: (a) Greater than 1 milliliter (mL) viable frozen bone marrow aspirated aliquot (preferred) collected in an ethylenediaminetetra-acetic acid (EDTA) tube, frozen, and stored at a temperature of -80 centigrade (°C), or; (b) Non-decalcified diagnostic bone marrow aspirate clot sections (block or slides) for MRD assessment: (i) A formalin fixed paraffin embedded (FFPE) block of bone marrow aspirate clot, or slides (preferably 5, if available), 5 micrometer each, of non-decalcified bone marrow, or; (ii) Slides (preferably 5, if available), bone marrow aspirate smear; (iii) Please note, bone marrow core sections are not acceptable samples for analysis; (iv) In exceptional circumstances when index myeloma clone cannot be identified from the archived bone marrow sample, a post-transplant sample can be used to identify myeloma clone with permission from the sponsor
* Must have residual disease as defined by detectable MRD (Adaptive Biotechnologies' NGS based MRD assay)
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2

Exclusion Criteria:

* A history of malignancy (other than multiple myeloma) unless all treatment of that malignancy was completed at least 2 years before consent and the participant has no evidence of disease before the of date of randomization. Exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years
* Must not have progressed on multiple myeloma (MM) therapy at any time prior to screening
* Have had prior treatment/therapy with: (a) Daratumumab or any other anti-cluster of differentiation 38 (CD38) therapies, (b) Focal radiation therapy within 14 days prior to randomization with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma. Radiotherapy within 14 days prior to randomization on measurable extramedullary plasmacytoma is not permitted even in the setting of palliation for symptomatic management, or (c) Plasmapheresis within 28 days of randomization
* Be exhibiting clinical signs of meningeal or central nervous system involvement due to multiple myeloma
* Have known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) less than (<) 50 percent (%) of predicted normal
* Have known moderate or severe persistent asthma within the past 2 years or current uncontrolled asthma of any classification
* Have any of the following: (a) Known history of seropositivity for human immunodeficiency virus (HIV); (b) Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]. Participants with resolved infection (that is, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR; (c) Seropositive for hepatitis C (anti-hepatitis C virus [HCV] antibody positive or HCV-RNA quantitation positive), except in the setting of a sustained virologic response, defined as aviremia at least 12 weeks after completion of antiviral therapy)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2026-05-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (73):
- United States (70):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, PC - HAL, Glendale, Arizona
  - Cancer Treatment Center of America Phoenix, Goodyear, Arizona
  - University of California San Diego (UCSD) - The Rebecca and John Moores Cancer Center, La Jolla, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Colorado Health, Fort Collins, Colorado
  - Yale University Medical Center, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University Cancer And Blood Center LLC, Athens, Georgia
  - Illinois Cancer Specialists, Niles, Illinois
  - Cancer Treatment Centers of America, Zion, Illinois
  - Fort Wayne Medical Oncology and Hematology American Oncology Partners, Fort Wayne, Indiana
  - Franciscan Health, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Cancer And Hematology Centers of Western Michigan PC, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - HCA MidAmerica Division Inc Research Medical Center, Kansas City, Missouri
  - Summit Medical Group/MD Anderson Cancer Center, Florham Park, New Jersey
  - Rutgers, The State Univ of NJ-Robert Wood Johnson Medical School-The Cancer Institute of NJ (CINJ), New Brunswick, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Northwell Health, Lake Success, New York
  - NYU Winthrop, Mineola, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Novant Oncology Research Institute, Winston-Salem, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Northwest Cancer Specialists PC, Portland, Oregon
  - Oregon Health And Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Reading Hospital/McGlinn Cancer Institute, West Reading, Pennsylvania
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Spartanburg Regional Health Services, Spartanburg, South Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology-Central South, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology P A, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center (UT Health San Antonio), San Antonio, Texas
  - Texas Oncology P A, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Cancer Center - Emily Couric Clinical Cancer Center - Women's Oncology Clinic, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - VA Puget Sound Healthcare System, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
- Canada (3):
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec Universite Laval Hopital de l Enfant Jesus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Badros A, Foster L, Anderson LD Jr, Chaulagain CP, Pettijohn E, Cowan AJ, Costello C, Larson S, Sborov DW, Shain KH, Silbermann R, Shah N, Chung A, Krevvata M, Pei H, Patel S, Khare V, Cortoos A, Carson R, Lin TS, Voorhees P. Daratumumab with lenalidomide as maintenance after transplant in newly diagnosed multiple myeloma: the AURIGA study. Blood. 2025 Jan 16;145(3):300-310. doi: 10.1182/blood.2024025746. PMID 39331724
- [Derived] Swan D, Henderson R, McEllistrim C, Naicker SD, Quinn J, Cahill MR, Mykytiv V, Lenihan E, Mulvaney E, Nolan M, Parker I, Natoni A, Lynch K, Ryan AE, Szegezdi E, Krawczyk J, Murphy P, O'Dwyer M. CyBorD-DARA in Newly Diagnosed Transplant-Eligible Multiple Myeloma: Results from the 16-BCNI-001/CTRIAL-IE 16-02 Study Show High Rates of MRD Negativity at End of Treatment. Clin Lymphoma Myeloma Leuk. 2022 Nov;22(11):847-852. doi: 10.1016/j.clml.2022.07.011. Epub 2022 Jul 21. PMID 35985959

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Currently, results posted till interim data cutoff date of 04-April-2024 (primary completion date).
Groups:
- Daratumumab + Lenalidomide: Participants received daratumumab 1800 milligrams (mg) subcutaneous (SC) injection weekly during Cycle 1 and Cycle 2 (that is, on Day 1, Day 8, Day 15 and Day 22 of each Cycle), followed by every-2-week dosing from Cycle 3 to Cycle 6 (that is, on Weeks 9, 11, 13, 15, 17, 19, and 21) and then every-4-week dosing from Cycle 7 onwards (that is, from Week 25). In addition, participants received maintenance therapy with lenalidomide 10 mg capsule orally (PO) from Day 1 to 28 in each treatment cycle. Participants received study treatment until confirmed disease progression (PD), unacceptable toxicity, or until end of study treatment, whichever occurred first. After Cycle 3, if lenalidomide was well tolerated, dose might be increased to 15 mg at the discretion of the investigator. Each treatment cycle was of 28 days.
- Lenalidomide: Participants received lenalidomide 10 mg capsule PO as maintenance therapy from Day 1 to Day 28 of each 28-day treatment cycle until confirmed PD, unacceptable toxicity, or the end of the study treatment, whichever occurred first. After Cycle 3, if lenalidomide was well tolerated, dose might be increased to 15 mg at the discretion of the investigator.
Period: Overall Study
Arm/Group | Daratumumab + Lenalidomide | Lenalidomide
Started | 99 | 101
Treated | 96 | 98
Completed | 5 | 10
Not Completed | 94 | 91
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 4 | 11
Not completed — Ongoing | 84 | 73
Not completed — Randomized but not treated | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daratumumab + Lenalidomide | Lenalidomide | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.12) | 60.8 (9.54) | 61 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 43 | 81
  Male | 61 | 58 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 81 | 89 | 170
  Unknown or Not Reported | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 1 | 6
  Black or African American | 20 | 24 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 67 | 68 | 135
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4
  Other | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 0 | 2
  United States | 97 | 101 | 198

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Minimal Residual Disease (MRD) Conversion From Baseline to 12 Months After Start of Maintenance Treatment as Determined by Next Generation Sequencing (NGS)
Description: Percentage of participants who achieved MRD negative (MRD conversion) status from baseline to 12 months after maintenance treatment was defined as percentage of participants who were MRD positive at baseline (randomization) and achieved MRD negative status (at 10^-5) during the time period from randomization to 12 months plus 2 months window, but prior to progressive disease (PD) and subsequent anti-myeloma therapy.
Time Frame: From randomization up to 12 months
Population: The full analysis set (FAS) which included all participants randomly assigned to daratumumab in combination with lenalidomide or the lenalidomide alone.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab + Lenalidomide | Lenalidomide
Number analyzed (Participants) | 99 | 101
percentage of participants | 50.5 [40.3 to 60.7] | 18.8 [11.7 to 27.8]
Statistical Analysis 1: Comparison: Daratumumab + Lenalidomide vs Lenalidomide; Test type: Superiority; p < 0.0001, stratified Cochran-Mantel-Haenszel (CMH) — Tested at 2-sided 0.05 significance level through stratified CMH method. Stratification factor included baseline cytogenetic risk per investigator'; Odds Ratio (OR) = 4.51, 95% CI 2-sided [2.37 to 8.57] — Odds ratio and 95% CI were estimated by Mantel-Haenszel method. Stratification factor included baseline cytogenetic risk per investigator's assessment (high risk versus standard/unknown risk) as used for randomization of the study

2. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: From randomization to either disease progression or death (up to 7.1 years)
Reporting Status: Not Posted, anticipated posting 2027-05

3. Secondary Outcome: Percentage of Participants Who Achieved Overall MRD (at 10^-5) Negativity Conversion From Baseline to End of Study Treatment Period
Time Frame: From randomization up to 30 days after last dose of study treatment or disease progression or initiation of subsequent therapy, whichever occurs first (up to 3 years)
Reporting Status: Not Posted, anticipated posting 2027-05

4. Secondary Outcome: Percentage of Participants Who Achieved Durable (Greater Than or Equal to [>=] 12 Months) MRD Negative Status (10^-5)
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2027-05

5. Secondary Outcome: Response Rates by International Myeloma Working Group (IMWG) 2016 Criteria
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2027-05

6. Secondary Outcome: Overall Survival (OS)
Time Frame: From randomization up to 7.1 years
Reporting Status: Not Posted, anticipated posting 2027-05

7. Secondary Outcome: Duration of Complete Response (CR)
Time Frame: From date of initial documentation of CR or sCR up to first documented disease progression or death due to disease progression whichever occurs first (up to 7.1 years)
Reporting Status: Not Posted, anticipated posting 2027-05

8. Secondary Outcome: Health-related Quality of Life: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-C30 (EORTC QLQ-C30)
Time Frame: From baseline (Cycle 1 Day 1) up to 7.1 years
Reporting Status: Not Posted, anticipated posting 2027-05

9. Secondary Outcome: Health-related Quality of Life: Change From Baseline in European Quality of Life Five Dimensions Questionnaire-5-level (EQ-5D-5L)
Time Frame: From baseline (Cycle 1 Day 1) up to 7.1 years
Reporting Status: Not Posted, anticipated posting 2027-05

10. Secondary Outcome: Health-related Quality of Life: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-Multiple Myeloma Module (EORTC QLQ-MY20)
Time Frame: From baseline (Cycle 1 Day 1) up to 7.1 years
Reporting Status: Not Posted, anticipated posting 2027-05

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: From Cycle 1 Day 1 up to 30 days after the last study treatment or day prior to start of subsequent antimyeloma therapy (up to 7.1 years)
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: From Cycle 1 Day 1 up to 30 days after the last study treatment or day prior to start of subsequent antimyeloma therapy (up to 4.9 years)
Description: Serious adverse events and Other adverse events were analyzed on safety analysis set which included all randomized participants who received at least 1 dose of study agent. All-cause mortality was assessed on all randomized participants.
Arm/Group | Daratumumab + Lenalidomide | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 5/99 | 9/101
Serious Adverse Events (participants affected / at risk) | 29/96 | 22/98
Other Adverse Events (participants affected / at risk) | 95/96 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab + Lenalidomide (N=96) | Lenalidomide (N=98)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Retinal Artery Embolism (Eye disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Complication Associated with Device (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0
Arthritis Infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 1 | 1
Covid-19 Pneumonia (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 2 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Escherichia Infection (Infections and infestations) | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Meningitis Cryptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 4
Pneumonia Legionella (Infections and infestations) | 1 | 0
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1 | 0
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Septic Shock (Infections and infestations) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-Cell Type Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Alcohol Abuse (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Melanocytic Hyperplasia (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab + Lenalidomide (N=96) | Lenalidomide (N=98)
Anaemia (Blood and lymphatic system disorders) | 21 | 17
Eosinophilia (Blood and lymphatic system disorders) | 3 | 2
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 25 | 28
Lymphopenia (Blood and lymphatic system disorders) | 23 | 13
Neutropenia (Blood and lymphatic system disorders) | 62 | 60
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 27
Atrial Fibrillation (Cardiac disorders) | 4 | 0
Atrial Flutter (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 4
Palpitations (Cardiac disorders) | 3 | 3
Sinus Bradycardia (Cardiac disorders) | 3 | 7
Sinus Tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 2
Ear Discomfort (Ear and labyrinth disorders) | 0 | 2
Ear Pain (Ear and labyrinth disorders) | 6 | 3
Hypoacusis (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 4
Androgen Deficiency (Endocrine disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1
Blepharitis (Eye disorders) | 0 | 3
Cataract (Eye disorders) | 4 | 1
Dry Eye (Eye disorders) | 2 | 3
Vision Blurred (Eye disorders) | 7 | 3
Visual Impairment (Eye disorders) | 2 | 1
Abdominal Distension (Gastrointestinal disorders) | 6 | 2
Abdominal Pain (Gastrointestinal disorders) | 17 | 11
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 2
Colitis (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 22 | 26
Dental Caries (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 59 | 54
Diverticulum (Gastrointestinal disorders) | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 13 | 5
Faeces Discoloured (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 4 | 3
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 4
Haematochezia (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 26 | 26
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 7 | 5
Toothache (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 17 | 11
Asthenia (General disorders) | 3 | 1
Chest Pain (General disorders) | 5 | 2
Chills (General disorders) | 6 | 4
Face Oedema (General disorders) | 2 | 2
Facial Pain (General disorders) | 2 | 1
Fatigue (General disorders) | 44 | 46
Gait Disturbance (General disorders) | 1 | 3
Generalised Oedema (General disorders) | 2 | 1
Influenza Like Illness (General disorders) | 12 | 14
Injection Site Bruising (General disorders) | 2 | 0
Injection Site Erythema (General disorders) | 6 | 1
Injection Site Pain (General disorders) | 2 | 0
Injection Site Reaction (General disorders) | 2 | 0
Localised Oedema (General disorders) | 2 | 1
Malaise (General disorders) | 3 | 2
Non-Cardiac Chest Pain (General disorders) | 7 | 7
Oedema Peripheral (General disorders) | 12 | 14
Pain (General disorders) | 2 | 1
Peripheral Swelling (General disorders) | 6 | 1
Pyrexia (General disorders) | 16 | 16
Temperature Intolerance (General disorders) | 5 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 8
Hypogammaglobulinaemia (Immune system disorders) | 9 | 0
Bronchitis (Infections and infestations) | 5 | 8
Cellulitis (Infections and infestations) | 2 | 2
Clostridium Difficile Infection (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 4 | 4
Covid-19 (Infections and infestations) | 27 | 26
Covid-19 Pneumonia (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 3 | 0
Ear Infection (Infections and infestations) | 2 | 0
Enterocolitis Infectious (Infections and infestations) | 2 | 0
Escherichia Infection (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 2 | 0
Herpes Zoster (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 1 | 5
Nasopharyngitis (Infections and infestations) | 8 | 2
Onychomycosis (Infections and infestations) | 2 | 0
Oral Candidiasis (Infections and infestations) | 0 | 2
Otitis Externa (Infections and infestations) | 1 | 2
Otitis Media (Infections and infestations) | 3 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 7 | 12
Rash Pustular (Infections and infestations) | 0 | 3
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 4
Rhinovirus Infection (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 8 | 9
Skin Infection (Infections and infestations) | 3 | 2
Tinea Pedis (Infections and infestations) | 3 | 0
Tooth Abscess (Infections and infestations) | 2 | 0
Tooth Infection (Infections and infestations) | 3 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 40 | 26
Urinary Tract Infection (Infections and infestations) | 10 | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 12 | 8
Epicondylitis (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 10
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 2
Limb Injury (Injury, poisoning and procedural complications) | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 2 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 2
Tooth Fracture (Injury, poisoning and procedural complications) | 2 | 3
Alanine Aminotransferase Increased (Investigations) | 16 | 13
Aspartate Aminotransferase Increased (Investigations) | 14 | 13
Blood Alkaline Phosphatase Increased (Investigations) | 7 | 8
Blood Bicarbonate Decreased (Investigations) | 1 | 2
Blood Creatinine Decreased (Investigations) | 0 | 2
Blood Creatinine Increased (Investigations) | 13 | 11
Blood Lactate Dehydrogenase Increased (Investigations) | 3 | 2
Blood Urea Increased (Investigations) | 2 | 0
Human Rhinovirus Test Positive (Investigations) | 2 | 0
Weight Decreased (Investigations) | 8 | 5
Weight Increased (Investigations) | 5 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 10 | 10
Dehydration (Metabolism and nutrition disorders) | 3 | 6
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 36
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 3
Polydipsia (Metabolism and nutrition disorders) | 2 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 2
Vitamin D Deficiency (Metabolism and nutrition disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 36
Back Pain (Musculoskeletal and connective tissue disorders) | 31 | 20
Bone Pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Flank Pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 22 | 21
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 9 | 8
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 10
Neck Pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 22 | 17
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 5 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Ageusia (Nervous system disorders) | 2 | 1
Amnesia (Nervous system disorders) | 2 | 0
Carotid Artery Stenosis (Nervous system disorders) | 2 | 0
Disturbance in Attention (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 18 | 16
Dysgeusia (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 24 | 17
Hypoaesthesia (Nervous system disorders) | 9 | 3
Memory Impairment (Nervous system disorders) | 4 | 2
Migraine (Nervous system disorders) | 2 | 3
Neuralgia (Nervous system disorders) | 4 | 2
Neuropathy Peripheral (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 7 | 9
Parosmia (Nervous system disorders) | 0 | 2
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 12 | 13
Syncope (Nervous system disorders) | 0 | 4
Tremor (Nervous system disorders) | 4 | 0
Affect Lability (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 6 | 3
Depression (Psychiatric disorders) | 7 | 7
Insomnia (Psychiatric disorders) | 15 | 8
Libido Decreased (Psychiatric disorders) | 2 | 0
Sleep Disorder (Psychiatric disorders) | 2 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 3 | 0
Pollakiuria (Renal and urinary disorders) | 5 | 1
Renal Cyst (Renal and urinary disorders) | 1 | 2
Renal Impairment (Renal and urinary disorders) | 3 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 2
Breast Pain (Reproductive system and breast disorders) | 2 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 5 | 2
Pelvic Pain (Reproductive system and breast disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 36
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 15
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 25 | 19
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 16 | 11
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 | 7
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 12 | 11
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 19 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 6
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 3 | 5
Pain of Skin (Skin and subcutaneous tissue disorders) | 2 | 0
Perioral Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 9
Rash (Skin and subcutaneous tissue disorders) | 9 | 12
Rash Erythematous (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 2 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 21 | 17
Rash Papular (Skin and subcutaneous tissue disorders) | 3 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 4 | 1
Sensitive Skin (Skin and subcutaneous tissue disorders) | 4 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 2 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1
Embolism Venous (Vascular disorders) | 2 | 3
Flushing (Vascular disorders) | 4 | 1
Hot Flush (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 14 | 10
Hypotension (Vascular disorders) | 6 | 6
Superficial Vein Thrombosis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT03901963/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT03901963/SAP_001.pdf